CLINICAL TRIAL: NCT05052411
Title: Beta Testing of a Smartphone App for HIV Prevention in Malaysian MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Malaya (Other); Yale University (Other)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21TW011665 (NIH)
Record Dates: First submitted 2021-08-25; First posted 2021-09-22 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: HIV Prevention Program
Keywords: PrEP; mHealth; mobile application

STUDY DESIGN:
Intervention Model Description: We will enroll 50 MSM for a total of 1 month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expanded beta testing of the JomPrEP app (Experimental): App usage assessments and analytics over a 1-month period.
  Interventions: Other: App usage assessments and analytics

INTERVENTIONS:
Other: App usage assessments and analytics — All participants will be given a brief overview of the purpose of the study followed by a survey on participant characteristics and barriers to accessing HIV testing and PrEP uptake and P/SUD support services. The participant will be observed downloading the JomPrEP app and instructed with a brief tutorial on the onboarding process. The participant will be told to keep the app for 1 month and encouraged to use all app components. At 30 days, the participant will complete a post-survey, to which the Systems Usability Scale will be added. App analytics will also be collected (e.g., the number of logins). Participants will be asked to provide feedback on functionality, performance, and errors encountered, motivation to use the app, overall experiences using the app, feedback for further refinement, and subjective impact of the app on HIV prevention.

SUMMARY:
This project will involve beta testing of the JomPrEP app to assess its usability and acceptability among Malaysian MSM.

DETAILED DESCRIPTION:
Given the evolving HIV epidemic among MSM and their challenges with accessing prevention services, we previously proposed to adapt, expand, and refine an existing app (namely the HealthMindr app) to deliver an integrated HIV prevention intervention that will promote HIV testing and linkage to PrEP and that incorporates screening and support for P/SUD for Malaysian MSM. We now plan to conduct expanded beta testing of the newly designed JomPrEP app to assess its usability and acceptability among Malaysian MSM.

Following wireframing and usability testing, Keymind (an experienced mobile app development company that has significant experience in building HIPAA-compliant apps, including HealthMindr) will apply a user interface (UI) design (i.e., colors/branding) to the interactive prototype, followed by the final development of the app (beta version). The objective of this study is to beta test this app to identify potential bugs and to ensure its usability in a real-world setting.

As part of the expanded beta testing, we will also evaluate the design, functionality, and usability of the JomPrEP app. This step is a critical stage of app development and will increase the ability of our research team to develop an acceptable and effective app.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative MSM
* Age more than or equal to 18
* Cis-gender men
* Condomless sex in the last 30 days
* Own a smartphone

Exclusion Criteria:

* Unable to provide informed consent
* Unable to read and understand English or Bahasa Malaysia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender men.
Enrollment: 50 (Actual)
Dates: Start 2022-03-13 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Usability of the JomPrEP app through the System Usability Scale | 1 month
  The Systems Usability Scale (SUS) will be used to assess the subjective usability of the app.
Usability of the JomPrEP app through app analytics | 1 month
  The investigators will collect app analytics, such as the number of log-ins to assess usability.
Usability of the JomPrEP app through app analytics | 1 month
  The investigators will collect app analytics, such as session duration to assess usability.
Usability of the JomPrEP app through app analytics | 1 month
  The investigators will collect app analytics, such as pages visited to assess usability.
Usability of the JomPrEP app through app analytics | 1 month
  The investigators will collect app analytics, such as frequency of use of app components to assess usability.
Usability of the JomPrEP app through app analytics | 1 month
  The investigators will collect app analytics, such as the duration of use of app components to assess usability.
Usability of the JomPrEP app through interviews | 1 month
  Participants will be asked to provide qualitative feedback on functionality, performance, and errors encountered, motivation to use the app, overall experiences using the app, feedback for further refinement, and subjective impact of the app on HIV prevention outcomes.
Acceptability of the JomPrEP app through the System Usability Scale | 1 month
  Point estimates for mean acceptability ≥50 for the System Usability Scale will be considered the minimum criteria for acceptability. The higher the score, the better the outcome. Minimum score for the scale is 0, maximum score is 100.
Acceptability of the JomPrEP app through calculated proportions | 1 month
  Proportion of participants accessing the app >0.60 will be considered the minimum criteria for acceptability.

SECONDARY OUTCOMES:
Feasibility of the JomPrEP app through the System Usability Scale | 1 month
  Point estimates for mean acceptability ≥50 for the System Usability Scale will be considered the minimum criteria for feasibility. The higher the score, the better the outcome. Minimum score for the scale is 0, highest score is 100.
Feasibility of the JomPrEP app through calculated proportions | 1 month
  Proportion accessing the app >0.60 will be considered the minimum criteria for feasibility.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Shrestha R, Altice FL, Khati A, Azwa I, Gautam K, Gupta S, Sullivan PS, Ni Z, Kamarulzaman A, Phiphatkunarnon P, Wickersham JA. Clinic-Integrated Smartphone App (JomPrEP) to Improve Uptake of HIV Testing and Pre-exposure Prophylaxis Among Men Who Have Sex With Men in Malaysia: Mixed Methods Evaluation of Usability and Acceptability. JMIR Mhealth Uhealth. 2023 Feb 16;11:e44468. doi: 10.2196/44468. PMID 36795465
- See also: Naeem F, Syed Y, Xiang S, et al. Development, Testing and Reporting of Mobile Apps for Psycho-social Interventions: Lessons from the Pharmaceuticals. Journal of Medical Diagnostic Methods. 2015;4(4). — https://www.longdom.org/open-access/development-testing-and-reporting-of-mobile-apps-for-psychosocialinterventions-lessons-from-the-pharmaceuticals-2168-9784-1000191.pdf
- See also: Bangor A, Kortum P, Miller J. Determining what individual SUS scores mean: adding an adjective rating scale. J. Usability Studies. 2009;4(3):114-123. — https://uxpajournal.org/determining-what-individual-sus-scores-mean-adding-an-adjective-rating-scale/
- See also: Brooke J, Jordan P, Thomas B, Weerdmeester B, McClelland I. Usability evaluation in industry. SUS: a'quick and dirty'usability scale. 1996:184-194. — https://www.routledge.com/Usability-Evaluation-In-Industry/Jordan-Thomas-McClelland-Weerdmeester/p/book/9780748404605